CLINICAL TRIAL: NCT05851677
Title: Disitamab Vedotin (RC48-ADC) in Patients With Breast Cancer: a Real-world Study
Brief Title: Disitamab Vedotin (RC48-ADC) in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Other Study IDs: LY2023-062-B
Record Dates: First submitted 2023-04-30; First posted 2023-05-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RC48-ADC: RC48-ADC for breast cancer
  Interventions: Drug: Disitamab vedotin

INTERVENTIONS:
Drug: Disitamab vedotin — recommended but not required regimen of 2.0mg/kg, iv, day1, every 2 weeks
  Other Names: RC48-ADC

SUMMARY:
To evaluate the efficacy and safety of Disitamab vedotin (RC48-ADC) in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer;
* Prior or current use of Disitamab vedotin (RC48-ADC);

Exclusion Criteria:

* Participating in clinical trials involving Disitamab vedotin (RC48-ADC) or not.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: breast cancer patients with prior or current use of Disitamab vedotin (RC48-ADC)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From the date of starting Disitamab vedotin to the date of first documentation of progression or death (up to approximately 1 years)
  The time from the date of starting Disitamab Vedotin to the date of disease progression as per RECIST version 1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse events | From the date of starting Disitamab vedotin to the end of the treatment (up to approximately 1 year)
  Adverse events during Disitamab Vedotin regimen will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital,School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No